CLINICAL TRIAL: NCT03615079
Title: Internet-based Cognitive Behavioral Therapy to Reduce Depressive Symptoms After Stroke Pilot/Feasibility Study
Brief Title: Internet-based CBT After Stroke Pilot
Acronym: iSAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Michael Mullen, Assistant Professor of Neurology, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 829426
Record Dates: First submitted 2018-06-18; First posted 2018-08-03 (Actual); Results first posted 2021-11-10 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Stroke; Depression
MeSH Terms: conditions — Stroke; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Behavioral Therapy (CBT) program (Other)
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — An 8-week, internet-based cognitive behavioral therapy (CBT) program for depression

SUMMARY:
Mood disorders occur in 25-30% of stroke patients and are associated with lower quality of life, higher mortality, increased healthcare utilization, and higher costs. Cognitive behavioral therapy (CBT) interventions have been shown to both treat and prevent post-stroke mood disorders, thus having the ability to improve quality of life and reduce costs. This study aims to test the feasibility of internet-based CBT combined with a telephone/email based coaching service after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age
* Acute ischemic stroke within the past 3 months
* Regular access to the internet, sufficient to allow a minimum of interactions with the internet daily, either through a personal smartphone or web-based internet browser.
* Subject is willing and able to participate in internet-based cognitive behavioral therapy
* Can participate in the program in English
* Willingness and ability to sign informed consent by the patient
* Symptoms of mild to moderately depressed mood, defined as a score of 5-19 on the Patient Health Questionnaire-9 at the time of study enrollment.

Exclusion Criteria:

* Severely depressed patients, defined by a score of 20+ on the Patient Health Questionnare-9 are excluded
* Patients with an active bipolar disorder diagnosis are excluded
* Patients with personality disorder diagnoses are excluded
* Patients with active suicidality or past suicide attempts are excluded
* History of schizophrenia or schizoaffective disorder
* Active participation in face-to-face psychotherapy prior to stroke
* Patients with a history of dementia are excluded
* Patients with aphasia, defined as a score of 1 or greater on NIH Stroke Scale Item 9 are excluded.
* Patients without regular internet access through a computer, tablet or smartphone are excluded.
* Subjects requiring long-term inpatient nursing care are excluded. For patients enrolled as inpatients, individuals being discharged to both home and acute rehab are eligible. Individuals being discharged to a skilled nursing facility or hospice are excluded.
* Expected life expectancy less than 6 months or other inability to comply with study follow-up.
* Pregnant women and prisoners are excluded

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mullen, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The proportion of subjects who engaged with the CBT application was not what was expected and as such enrollment was expanded with the goal of getting 20 subjects to use the application.
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy (CBT) Program
Started | 28
Completed | 11
Not Completed | 17

BASELINE CHARACTERISTICS:
Population: Subjects who engaged with the CBT application at least once
Arm/Group | Cognitive Behavioral Therapy (CBT) Program
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Depressive Symptoms Over Time
Description: Subject's depressive symptoms will be quantified using the Patient Health Questionnaire 9. This assessment includes 9 close-ended questions with a scoring system ranging from 0 to 27. Scores greater than 10 are considered "positive" for depressive symptoms. We will compare the average PHQ-9 score at study enrollment to the PHQ-9 at 90 days to determine the reduction in depressive symptoms over time.
Time Frame: Baseline and 90 days
Population: 1 subject missing day 90 PHQ-9
Measure: Median (Inter-Quartile Range); unit: scores on scale
Arm/Group | Cognitive Behavioral Therapy (CBT) Program
Number analyzed (Participants) | 10
scores on scale | 6 [5 to 7]

2. Secondary Outcome: Quality of Life Assessed by the EuroQOL-5D
Description: EuroQOL-5D questionnaire that measures health related quality of life. The scale ranges from 1 to 100, with higher scores indicating better outcomes.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Cognitive Behavioral Therapy (CBT) Program
Number analyzed (Participants) | 11
scores on a scale | 73 (16)

ADVERSE EVENTS:
Time Frame: 90 days
Description: Definition did not differ
Arm/Group | Cognitive Behavioral Therapy (CBT) Program
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

LIMITATIONS AND CAVEATS:
The aim of this study was to enroll 20 subjects into the computer based cognitive-behavioral therapy intervention. Unfortunately enrollment was slower than expected and the proportion of enrolled subjects who utilized the application was low, limiting the analysis and preventing meaningful conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT03615079/Prot_SAP_000.pdf